CLINICAL TRIAL: NCT05436756
Title: Chronic Post-leptospirosis Manifestations in Reunion
Acronym: LEPTONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/CHU/16
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Leptospirosis
MeSH Terms: conditions — Leptospirosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sampling and clinical data collection (Other): * Biological sampling and collection:
    * whole blood: 1 dry tube for IgG and IgM anti-leptospirosis serology (volume depending on the patient's weight)
    * urine: 1 bottle of 30ml
  * Freezing of serum after centrifugation
  * Storage at Biological Ressources Center
  * Collection of clinico-biological data on a dedicated eCRF
  Interventions: Other: Biological sampling and collection

INTERVENTIONS:
Other: Biological sampling and collection — * Biological sampling and collection:
    * whole blood: 1 dry tube for IgG and IgM anti-leptospirosis serology (volume depending on the patient's weight)
    * urine: 1 bottle of 30ml
  * Freezing of serum after centrifugation
  * Storage
  * Collection of clinico-biological data on a dedicated eCRF

SUMMARY:
Leptospirosis is a zoonosis caused by spirochetes, pathogenic bacteria of the genus Leptospira. It is transmitted to humans through mucocutaneous lesions by contact with water or soil contaminated by the urine of animal reservoirs (rats, dogs, pigs, cattle, etc.). Exposure to fresh water, contact with water or soil contaminated with animal waste are the main risk factors.

This disease is an important public health problem in humans and animals. The annual global incidence is estimated at nearly one million cases with a mortality of 5 to 10% for all cases combined and up to 50% in the event of multi-organ failure. The number of cases is growing and the disease is probably more widespread because it is underdiagnosed. The incidence could increase further in the coming decades due to climate change and rapid urbanization.

In the Overseas Departments and Regions (DROM), it is an endemic condition and its incidence is 10 to 100 times higher than that of mainland France, mainly for climatic reasons. In Réunion, the disease is notifiable with a number of notified cases ranging from 70 to more than 100 cases per year in recent years. Nearly 90% of confirmed cases were hospitalized and more than a third of patients stayed in intensive care.

Recently, a multicenter cohort of patients hospitalized with leptospirosis in La Réunion (COLEPT) was funded by Inserm to identify the severity factors of the disease in patients hospitalized in one of the 4 hospitals on the island. A community of hospital practitioners active on this theme has been identified and constitutes the core of this project. The main objective of the study, the inclusions of which began in January 2020, is to identify the severity factors of leptospirosis in Reunion. Patient follow-up is planned for up to 1 year with 2 medical visits at 1 month and 1 year and 2 telephone interviews on quality of life.

The disease is generally perceived as a purely acute condition with a rapid ad integrum recovery. Nevertheless, the evolution at a distance has been little evaluated. A few publications report complications and elements of chronicity in the medium/long term (>1 year) which would require monitoring these patients over a longer period. Regarding these potential chronic manifestations, they may be chronic fatigue, uveitis, renal failure, chronic renal carriage with urinary excretion of leptospires, myalgia and muscle weakness, headaches, malaise but also cardiac or neurological manifestations. A Dutch study conducted on subjects with confirmed diagnosis reported 30% of patients with chronic post-leptospirosis symptoms which persisted in 21% of subjects more than 24 months after infection, but very few data are available on the chronic forms.

The objective will be to study the future of patients beyond 1 year of infection in clinical and serological terms, but also in terms of quality of life, use of alternative medicines and complementary and health literacy profiles.

ELIGIBILITY:
Inclusion Criteria:

* Adult or child subjects having been included in the COLEPT cohort with confirmed leptospirosis Where
* Adult subjects or children hospitalized for leptospirosis confirmed within 12-18 months before LEPTONIC inclusion;
* Be resident in Reunion
* Ability to answer a telephone questionnaire
* Benefit from a social security scheme

Exclusion Criteria:

* Refusal of participation by the patient or his entourage if the patient is physically unable to give his opinion (coma, resuscitation, etc.).
* Exclusion or premature termination of participation in the COLEPT cohort
* Patient under judicial safeguard, guardianship or curatorship, under activated future protection mandate and family authorization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-07-24 (Estimated); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with chronic post-leptospirosis symptom(s) persisting 2 years after infection. | two years

CONTACTS AND LOCATIONS:
Locations (4):
- France (2):
  - CHOR, Saint-Paul
  - DIALLO, Saint-Pierre
- Reunion (2):
  - GHER, Saint-Benoît
  - CHU de la Réunion, Saint-Denis

IPD SHARING:
Plan to Share IPD: No